CLINICAL TRIAL: NCT05984927
Title: A Phase 1/2a Open-label Study to Evaluate Safety, Tolerability and Preliminary Efficacy of NG101 AAV Gene Therapy in Subjects With Wet Age-Related Macular Degeneration
Brief Title: NG101 AAV Gene Therapy in Subjects With Wet Age-Related Macular Degeneration
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Elisigen, Inc. (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NG101WA-01
Record Dates: First submitted 2023-07-24; First posted 2023-08-09 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Age-Related Macular Degeneration
Keywords: Wet macular degeneration; Neovascular Age-Related Macular Degeneration; Macular Degeneration; Choroidal Neovascularization; Retinal Degeneration; Eye Diseases; Retinal Diseases; Angiogenesis Inhibitors; Angiogenesis Modulating Agents; Growth Substances; Growth Inhibitors; Antineoplastic Agents; Gene Therapy; Anti-vascular endothelial growth factor therapy; Anti-VEGF therapy
MeSH Terms: conditions — Macular Degeneration; Wet Macular Degeneration; Choroidal Neovascularization; Retinal Degeneration; Eye Diseases; Retinal Diseases

STUDY DESIGN:
Intervention Model Description: Dose Escalation Study with 3 dose cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- NG101 Gene Therapy Group 1 (Experimental): Single subretinal injection of 1x10^9 vector genomes of NG101 AAV gene therapy
  Interventions: Genetic: NG101 AAV gene therapy
- NG101 Gene Therapy Group 2 (Experimental): Single subretinal injection of 3x10^9 vector genomes of NG101 AAV gene therapy
  Interventions: Genetic: NG101 AAV gene therapy
- NG101 Gene Therapy Group 3 (Experimental): Single subretinal injection of 8x10^9 vector genomes of NG101 AAV gene therapy
  Interventions: Genetic: NG101 AAV gene therapy

INTERVENTIONS:
Genetic: NG101 AAV gene therapy — Sub retinal injection of NG101 (a non-replicating adeno-associated virus serotype 8 (AAV8) vector
  Other Names: NG101

SUMMARY:
This study will evaluate the safety, tolerability, and preliminary efficacy of NG101 AAV gene therapy administered by subretinal injections into a single selected eye as a single selected dose for patients with wet age-related macular degeneration (wAMD).

DETAILED DESCRIPTION:
This is a Phase 1/2a, multicenter, open-label, dose escalation study to evaluate the safety, tolerability, and preliminary efficacy of NG101 AAV gene therapy, administered by subretinal injection in patients with active wAMD symptoms. The study will be conducted at approximately 5 sites in Canada and the USA.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥ 50 and ≤ 89 years of age with a diagnosis of active subfoveal CNV secondary to wAMD in the Study Eye
2. BCVA between 20/40 and 20/400 in the Study Eye, with BCVA decrement primarily attributable to wAMD
3. Administration of at least 3 anti-VEGF (vascular endothelial growth factor) injections in the study eye in the past 6 months for clinically active wAMD, the most recent of which was within 1 month prior to Screening Day -14 (Visit 1).
4. Must be pseudo phakic (status post cataract surgery) in the Study Eye
5. Female and Male reproductive status: Female subjects must be either: (1) of non-childbearing potential; or (2) of childbearing potential and using an acceptable method of birth control with a negative pregnancy test. Male subjects agree to refrain from sperm donations and practice contraception to avoid any pregnancy for 3 months after administration of NG101.
6. Normal blood pressure (BP) and heart rate (HR), or near normal BP and HR not considered clinically significant (NCS) by the Investigator at the Screening Day -14 (Visit 1) and Day -7 (Visit 2)
7. Willing and able to provide written, signed informed consent after the nature of the study has been explained and prior to the performance of any study-related procedures
8. Willingness and ability to comply with schedule for follow-up visits and postoperative evaluations

Exclusion Criteria:

1. CNV or macular edema in the Study Eye secondary to any causes other than AMD
2. Any condition preventing visual acuity improvement in the Study Eye, e.g., fibrosis, atrophy, or retinal pigment epithelial tear involving the center of the macula
3. Any ophthalmic condition that precludes adequate ophthalmic examination or requires treatment
4. Retinal detachment or history of retinal detachment in the Study Eye
5. Active uncontrolled glaucoma with intraocular pressure (IOP) ≥ 30 mmHg despite treatment with more than 2 glaucoma medications, advanced glaucoma with cup-to-disc ratio of ≥ 0.9, visual field defects secondary to glaucoma that involve the macula, and/or optic atrophy from glaucoma
6. History of intravitreal therapy in the Study Eye, such as intravitreal steroid injection or an investigational product, other than anti-VEGF therapy, in the 6 months prior to Screening
7. History of vitrectomy, trabeculectomy, glaucoma tube-shunt procedure, minimally invasive glaucoma surgery (MIGS) device, or other filtration surgery in the Study Eye
8. Photodynamic therapy or retinal laser for the treatment of wAMD within the last 6 months
9. Any prior therapeutic radiation in the region of the Study Eye such as whole brain radiation, proton beam radiation, gamma knife treatment, or plaque brachytherapy
10. Any previous intraocular or refractive surgery on the Study Eye within 6 months
11. Any previous gene therapy in the Study Eye
12. Presence of an ocular implant in the Study Eye at Screening, excluding intraocular lens and custom flex iris prosthesis
13. Any diabetic retinopathy or other retinal vascular disease including retinal vein occlusion, retinal artery occlusion, retinal arterial macro aneurysm, ocular ischemic syndrome, retinal vasculitis, vitritis, posterior uveitis
14. Medically uncontrolled diabetes, defined as HbA1C > 8.0
15. History of ocular melanoma
16. History of any known inherited retinal disease
17. Currently taking any anticoagulant therapy, which is deemed medically necessary and cannot be permanently stopped at least 2 weeks prior to NG101 injection, excluding prophylactic low-dose aspirin therapy
18. Any underlying systemic diseases as unstable or severe cardiovascular, cerebrovascular, dementia or neurodegenerative diseases of a level that prevents adequate evaluation of the subject during the study, active malignancy or currently undergoing treatment for active malignancy at Screening or a history of malignancy that precludes completion of this 260 week study, and immunocompromised conditions and/or need for immunosuppressive therapy
19. Active hepatitis B or C
20. History of human immunodeficiency virus (HIV), active tuberculosis, and/or syphilis
21. Any significant illness that would preclude study compliance and follow-up
22. Subjects who, in the Investigator's opinion, lack the mental capacity to provide written informed consent for study participation

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | From Day 0 (pre-treatment) through Week 24
  Incidence and severity of ocular and non-ocular adverse events (AEs) for each cohort

SECONDARY OUTCOMES:
Ocular and Non -Ocular Adverse Events after week 24 | From Day 0 (pre-treatment) and through Weeks 52, 104, 156, 208 and 260
  Incidence and severity of ocular and non-ocular AEs from Day 0 (pre-treatment) through Weeks 52 and Week 260 for each cohort
Systemic Immunogenic Response | From Day -14 to Weeks 4, 8, 12, 24, 52, and 104
  Change in concentration of Anti-NG101 Transgene protein (aflibercept) antibodies, Anti-AAV8 Neutralizing antibodies, and Anti-AAV8 Antibodies in serum samples
Systemic Immunogenic Response | From Day -14 to Weeks 4, 12, and 104
  Change in concentration of expressed aflibercept protein in serum samples
Systemic Immunogenic Response | From Day -14 to Day 7, and Weeks 2, 4, and week 12.
  Change in AAV vector (NG101) genome copies as measured by qPCR (quantitative polymerase chain reaction) in blood samples
Systemic Immunogenic Response | From Day 0 (pre-treatment) to Weeks 24, 52, and 104
  Change in concentration of expressed aflibercept protein in vitreous samples
Signs of CNV (choroidal neovascularization) Activity | From Day -7 to Weeks 8, 24, 52, and 104
  Change of 1 or more signs of CNV activity assessed by OCT (Optical coherence tomography)
Central Subfield Thickness (CST) | From Day -7 to Weeks 24, 52, 104, 156, 208, and 260
  Change in CST assessed with OCT
Best Corrected Visual Acuity (BCVA) | From Day -7 to Weeks 24, 52, 104, 156, 208 and 260
  Change in BCVA assessed with Early Treatment Diabetic Retinopathy Study (ETDRS) scale
Cumulative Number of Rescue Therapy Injections | Through Weeks 24, 52, 104, 156, 208, and 260
  The cumulative number of rescue therapy injections per subject to maintain CNV control in the Study Eye

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Riemann, MD, Principal Investigator — Neuracle Genetics, Inc. Medical Director
Locations (5):
- United States (2):
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Retina Consultants of Texas, Bellaire, Texas
- Canada (3):
  - Vancouver Coastal Health Research Institute, Vancouver, British Columbia
  - Sunnybrook Ophthalmology and Vision Services, Toronto, Ontario
  - Vitreous Retina Macula Specialists of Toronto, Toronto, Ontario